CLINICAL TRIAL: NCT05775406
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Intravenously Administered KT-253 in Adult Patients with High Grade Myeloid Malignancies and Acute Lymphocytic Leukemia, Lymphoma, and Advanced Solid Tumors
Brief Title: Safety and Clinical Activity of KT-253 in Adult Patients with High Grade Myeloid Malignancies, Acute Lymphocytic Leukemia, Lymphoma, Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT253-AL-101
Record Dates: First submitted 2023-02-10; First posted 2023-03-20 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Myeloid Malignancies; Acute Lymphocytic Leukemia; Lymphomas; Advanced Solid Tumors
Keywords: KT-253; MDM2; High Grade MDS/MPN; ALL; AML; Lymphoma; Solid tumor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 Dose Escalation Arm A in patients with R/R Solid Tumors and Lymphomas (Experimental): KT-253 dosed intravenous (IV) once every three weeks in 21-day cycles
  Interventions: Drug: KT-253
- Phase 1 Dose Escalation Arm B in patients with R/R High Grade Myeloid Malignancies and ALL (Experimental): KT-253 dosed IV once every three weeks in 21-day cycles
  Interventions: Drug: KT-253

INTERVENTIONS:
Drug: KT-253 — KT-253 will be administered intravenously per the defined protocol frequency and dose level.

SUMMARY:
This Phase 1 study will evaluate the safety, tolerability, pharmacokinetics/pharmacodynamics (PK/PD), and clinical activity of KT-253 in adult patients with relapsed or refractory (R/R) high grade myeloid malignancies, acute lymphocytic leukemia (ALL), R/R lymphoma, myelofibrosis, and R/R solid tumors. The study will identify the pharmacologically optimal dose(s) (MTD) of KT-253 as the recommended Phase 2 dose (RP2D), based on all safety, PK, PD, and efficacy data.

DETAILED DESCRIPTION:
This is an open-label Phase 1 (dose escalation) first-in-human study (FIH) of KT-253 in adult patients. This study will be initiated in patients with lymphomas, and solid tumors and then subsequently in patients with advanced high grade myeloid malignancies and ALL. Therefore, the study is comprised of two arms to characterize the safety and tolerability of ascending doses of KT-253 in each arm. Arm A will consist of patients with lymphomas and advanced solid tumors and Arm B will consist of patients with high grade myeloid malignancies and ALL.

ELIGIBILITY:
Inclusion Criteria:

1. All Participants:

   * Eastern Cooperative Oncology Group performance status: 0-2.
   * Resolved acute effects of any prior therapy except for alopecia to baseline severity or Grade ≤1 NCI CTCAE and Grade ≤2 neuropathy
   * Adequate organ function at screening
2. Solid Tumors and Lymphoma (Arm A) ONLY

   * Histologically or pathologically confirmed solid tumor or lymphoma.
   * Relapsed and/or refractory (R/R) disease to at least two prior standard-of-care treatments or tumors for whom standard therapies are not available.
3. Advanced high grade myeloid malignancies, and Acute Lymphocytic Leukemia (Arm B) ONLY • Primary diagnosis of AML, ALL, High/Very High-risk MDS, MDS/MPN. Must be relapsed/refractory to standard therapies.

Exclusion Criteria:

1. All Participants:

   * Ongoing unstable cardiovascular function.
   * Major surgery requiring general anesthesia within 4 weeks prior to first dose of study drug.
   * History of or active concurrent malignancy unless disease-free for ≥ 2 years.
   * Known presence of p53 mutations in tumor tissue or blood, which are known to completely inactivate p53 transcriptional activity
2. Solid Tumors and Lymphoma (Arm A) ONLY

   * Known active uncontrolled or symptomatic central nervous system (CNS) metastases.
   * Autologous or allogenic hematopoietic stem cell transplant (HSCT) within six months prior to first dose of study drug or participant has progressed within six months from the day of stem cell infusion (for lymphoma participants only).
   * Exposures to anticancer therapy or investigational therapy within 2 weeks or 5 half-lives whichever is longer prior to the first dose of study drug.
   * Received immunotherapy/biologic treatment or investigational therapy within 4 weeks prior to first dose of KT-253, including tumor vaccines and checkpoint inhibitors.
3. Advanced high grade myeloid malignancies, and Acute Lymphocytic Leukemia (Arm B) ONLY

   * Active CNS leukemia. Participants with symptoms suggestive of CNS disease will require a lumbar puncture to rule out CNS disease.
   * Prior chemotherapy/radiation (including craniospinal radiation) within 2 weeks prior to the first dose of study drug.
   * Received allogeneic hematopoietic cell transplantation (HCT) <12 weeks prior to first dose or donor lymphocyte infusion (DLI) without conditioning <4 weeks prior to first dose.
   * Received autologous stem cell transplant (ASCT) < 4 weeks prior to first dose or the patient has not recovered from transplant associated toxicities to ≤ grade 1 prior to the first dose of study drug.
   * Received chimeric antigen receptor therapy or other modified T cell therapy <3 weeks prior to the first dose.
   * Patients with signs or symptoms of Grade ≥ 2 acute or chronic graft versus host disease (GVHD) within 2 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | From the time of signing ICF through 30 days after last dose of study drug or prior to start of a new anticancer therapy
  Adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0
Maximum Tolerated Dose (MTD) and recommended Phase 2 dose (RP2D) in Patients | From the time of the first dose of study drug through 30 days after the last dose of study drug or prior to start of a new anticancer therapy
  MTD and RP2D will be determined in patients with R/R high grade myeloid malignancies, ALL, and separately, in patients with lymphomas and advanced solid tumors

SECONDARY OUTCOMES:
Area under the Plasma Concentration versus Time Curve (AUC) of KT-253 | Blood samples for PK analysis collected up to Day15 during cycle 1 and cycle 2 (each cycle is 21 days)
  To determine the AUC from plasma concentrations in patients
Maximum Plasma Concentration of KT-253 (Cmax) | Blood samples for PK analysis collected up to Day15 during cycle 1 and cycle 2 (each cycle is 21 days)
  To determine the Cmax from plasma concentrations in patients
Time to maximum plasma concentration of KT-253 (Tmax) | Blood samples for PK analysis collected up to Day15 during cycle 1 and cycle 2 (each cycle is 21 days)
  To determine the Tmax from plasma concentrations in patients
Evidence of Clinical Activity of KT-253 in AML patients | From the time of the first dose of study drug through 30 days after the last dose of study drug or until disease recurrence or death, whichever occurs first, about 18 months
  Percentage of patients with Morphologic leukemia free state (MLFS), complete remission (CR), CR with partial hematologic recovery (CRh) according to the European LeukemiaNet (ELN) response criteria.
Evidence of Clinical Activity of KT-253 in ALL patients | From the time of the first dose of study drug through 30 days after the last dose of study drug or until disease recurrence or death, whichever occurs first, about 18 months
  Hematological remission rate defined as CR and CRh per NCCN guidelines
Evidence of Clinical Activity of KT-253 in High/Very High-Risk Myelodysplastic syndromes (MDS) patients | From the time of the first dose of study drug through 30 days after the last dose of study drug or until disease recurrence or death, whichever occurs first, about 18 months
  CR or CR equivalent, partial remission (PR),CR with limited count recovery, CRh, and hematologic improvement (HI) per revised International Working Group (IWG) criteria
Evidence of Clinical Activity of KT-253 in MDS/ Myeloproliferative Neoplasms (MPN) patients | From the time of the first dose of study drug through 30 days after the last dose of study drug or until disease recurrence or death, whichever occurs first, about 18 months
  Percentage of patients with CR, PR, and Marrow Response per MDS/MPN IWG
Evidence of Clinical Activity of KT-253 in R/R Lymphoma patients | From Baseline scan until first documented progression or death from any cause, whichever comes first , about 18 months
  Overall Response Rate (ORR) based on Investigator's assessment as per Lugano criteria 2014 for Lymphomas
Evidence of Clinical Activity of KT-253 in R/R Solid Tumor patients | From Baseline scan until first documented progression or death from any cause, whichever comes first, about 18 months
  Overall Response Rate (ORR) defined as percentage of patients with Complete Response or Partial Response per RECIST 1.1
Duration of Response (DoR) in Patients Treated with KT-253 | From date of first of response to the date of documented first progression or death whichever comes first, about 18 months
  Duration of Response (DoR) in R/R high grade myeloid malignancies and ALL, R/R lymphoma and R/R solid tumor patients treated with KT-253

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Gollerkeri, MD, Study Director — Kymera Therapeutics, Inc.
Locations (11):
- United States (11):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No